CLINICAL TRIAL: NCT01670110
Title: A Randomized, Placebo Controlled Clinical Trial of SOM230 (Pasireotide LAR) In Severe Polycystic Liver Disease
Brief Title: Pasireotide LAR in Severe Polycystic Liver Disease
Acronym: SOM230
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Marie Hogan, Assistant Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 11-007405
Record Dates: First submitted 2012-08-17; First posted 2012-08-21 (Estimated); Results first posted 2020-03-02 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Somatostatin Analogs; Polycystic Liver Disease; Autosomal Dominant Polycystic Kidney Disease; Autosomal Dominant Polycystic Liver Disease
Keywords: Polycystic Liver Disease; Autosomal dominant polycystic kidney disease; Autosomal dominant polycystic liver disease; Somatostatin analogs; Pasireotide LAR; SOM230
MeSH Terms: conditions — Polycystic liver disease; Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pasireotide LAR (SOM230) (Active Comparator): Active Pasireotide LAR
  Interventions: Drug: Pasireotide LAR
- placebo injection (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pasireotide LAR — Injectible, 60mg per month
  Arms: Pasireotide LAR (SOM230)
Drug: Placebo — To be injected once per month
  Arms: placebo injection

SUMMARY:
The purpose of this study is to compare SOM230 treatment to placebo. The investigators will also assess the efficacy and safety of SOM230 in reducing total liver volume and improving quality of life.

DETAILED DESCRIPTION:
Pasireotide (SOM230) is a novel multi-receptor-targeted analog that has high affinity for four of the five SST receptor subtypes (SSTr1, SSTr2, SSTr3 and SSTr5); it has a 40-fold higher affinity and 158-fold higher functional activity for the SST5 receptor than octreotide. Because of its broad receptor binding profile, pasireotide may be more potent in Polycystic Liver Disease (PLD) than octreotide. In this randomized double blind placebo controlled trial the investigators will compare SOM230 treatment to placebo for 12 months in patients with PLD. The primary endpoints will be assessed at 12 months and patients receiving placebo then crossed over to SOM230, permitting all participants to receive SOM230 for the subsequent two years. Magnetic resonance imaging (MRI) will be used to assess liver volume - the primary endpoint, which will be assessed at baseline, end of years 1 and 3. This study will assess the efficacy and safety of SOM230 in reducing total liver volume and improving quality of life over 12 months. (The investigators will not be assessing efficacy at 24 months.) The therapy way be effective in PLD but also may prove to be effective for many more patients with Polycystic Kidney Disease (PKD) which will be evaluated using eGFR and kidney volume using MRI.

The investigators plan to add other sub-sites in other locations.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Age ≥ 18 years.
* Diagnosis of PLD associated with ADPKD (meeting the Modified Ravine's criteria) or isolated ADPLD (defined by the criteria described by Reynolds et al)
* Severe PLD defined as a liver volume >4000mL or symptomatic disease due to mass effects from hepatic cysts (must be able to undergo MRI or CT scan to determine this).
* Not a candidate for or declining surgical intervention.
* Capable of providing informed consent.
* Life expectancy ≥ 12 weeks
* Patients with a known history of impaired fasting blood glucose (glucose >100 and <126) may be included at the discretion of the PI. These patients should be monitored closely throughout the trial and antihyperglycemic treatment adjusted as necessary. Patients that are deemed non eligible due to elevated glucose can be re-screened after adequate medical treatment.
* Adequate end organ function as defined by:
* Adequate bone marrow function:

  * WBC ≥ 2.5 x 109/L
  * Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L
  * Platelets ≥ 100 x 109/L
  * Hb ≥ 9 g/dL
* No evidence of significant liver disease:

  * Serum bilirubin ≤1.5 x ULN
  * INR < 1.3
  * ALT and AST ≤ 2 x ULN
* Estimated glomerular filtration rate (eGFR) >30 ml/min/m2
* Serum amylase and lipase ≤ 1.5 x ULN
* Alkaline phosphatase ≤ 2.5 x ULN
* Written informed consent obtained prior to any screening procedures
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures

Exclusion Criteria:

* Patients will be considered ineligible for this study if they meet any of the following criteria:
* Patients with a known hypersensitivity to SST analogs or any component of the pasireotide LAR or SQ formulations.
* Patients with known malabsorption syndrome, short bowel or chologenic diarrhea not controlled by specific therapeutic means.
* Patients with abnormal coagulation (PT or a PTT elevated by 30% above normal limits).
* Patients on continuous anticoagulation therapy. Patients who were on anticoagulant therapy must complete a washout period of at least 10 days and have confirmed normal coagulation parameters before study inclusion.
* Patients with symptomatic cholelithiasis.
* Patients who are not biochemically euthyroid.
* Patients with known history of hypothyroidism are eligible if they are on adequate and stable re-placement thyroid hormone therapy for at least 3 months.
* Serum magnesium ≥ ULN
* QT-related exclusion criteria:
* QTcF at screening > 470 msec
* Patients with a history of syncope or family history of idiopathic sudden death
* Patients who have sustained or clinically significant cardiac arrhythmias
* Risk factors for Torsades de Pointes such as hypokalemia, hypomagnesemia, cardiac failure, clinically significant/symptomatic bradycardia, or high-grade AV block
* Patients with concomitant disease(s) that could prolong QT such as autonomic neuropathy (caused by diabetes, or Parkinson's disease), HIV, cirrhosis, uncontrolled hypothyroidism or cardiac failure
* Family history of long QT syndrome
* Concomitant medications known to prolong the QT interval.
* Potassium < or = to 3.5
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:
* Patients who have Uncontrolled diabetes as defined by HbA1c>8%* despite adequate therapy
* Patients with the presence of active or suspected acute or chronic uncontrolled infection or with a history of immunodeficiency, including a positive HIV test result (ELISA and Western blot). An HIV test will not be required; however, previous medical history will be reviewed.
* Non-malignant medical illnesses that are uncontrolled or whose control may be jeopardized by the treatment with this study treatment.
* Liver disease such as cirrhosis, decompensated liver disease, chronic active hepatitis or chronic persistent hepatitis.
* Baseline ALT or AST >3x ULN
* Patients with life-threatening autoimmune and ischemic disorders.
* Uncontrolled hypertension
* Patients who have a history of a primary malignancy, with the exception of locally excised non-melanoma skin cancer and carcinoma in situ of uterine cervix. (Patients who have had no evidence of disease from primary cancer for 3 or more years are allowed to participate in the study.)
* History of pancreatitis
* Patients with a known history of hepatitis B or C
* Presence of Hepatitis B surface antigen (HbsAg)
* Presence of Hepatitis C antibody (anti-HCV)
* Patients with a history of, or current, alcohol misuse/abuse within the past 12 months
* Known gallbladder or bile duct disease, acute or chronic pancreatitis
* Patients who have any current or prior medical condition that may interfere with the conduct of the study or the evaluation of its results in the opinion of the Investigator or the Sponsor's Medical Monitor
* Use of an investigational drug within 1 month prior to dosing
* Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will not be able to complete the entire study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie C Hogan, MD PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Hogan MC, Chamberlin JA, Vaughan LE, Waits AL, Banks C, Leistikow K, Oftsie T, Madsen C, Edwards M, Glockner J, Kremers WK, Harris PC, LaRusso NF, Torres VE, Masyuk TV. Pansomatostatin Agonist Pasireotide Long-Acting Release for Patients with Autosomal Dominant Polycystic Kidney or Liver Disease with Severe Liver Involvement: A Randomized Clinical Trial. Clin J Am Soc Nephrol. 2020 Sep 7;15(9):1267-1278. doi: 10.2215/CJN.13661119. Epub 2020 Aug 25. PMID 32843370
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pasireotide LAR (SOM230) | Placebo Injection
Started | 33 | 15
Completed | 29 | 12
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pasireotide LAR (SOM230) | Placebo Injection | Total
Number analyzed (Participants) | 33 | 15 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.16 (8.63) | 51.40 (7.97) | 50.55 (8.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 12 | 43
  Male | 2 | 3 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 29 | 15 | 44
  African American | 1 | 0 | 1
  Other | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 33 | 15 | 48

OUTCOME MEASURES:

1. Primary Outcome: Change in Liver Volume
Description: Percent change was calculated for liver volumes using the equation=[(12 month value-baseline value)/baseline value]*100*12/12 month
Time Frame: baseline , 12 month
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Pasireotide LAR (SOM230) | Placebo Injection
Number analyzed (Participants) | 29 | 12
percentage of change | -3.36 (7.33) | 6.29 (6.97)
Statistical Analysis 1: Comparison: Pasireotide LAR (SOM230) vs Placebo Injection; Test type: Superiority; p = 0.001, ANCOVA

2. Primary Outcome: Change in Kidney Volume
Description: Percent change was calculated for kidney volumes using the equation=[(12 month value-baseline value)/baseline value]*100*12/12 month
Time Frame: baseline to 12 months
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Pasireotide LAR (SOM230) | Placebo Injection
Number analyzed (Participants) | 29 | 12
percentage of change | -1.37 (3.52) | 3.85 (4.49)
Statistical Analysis 1: Comparison: Pasireotide LAR (SOM230) vs Placebo Injection; Test type: Superiority; p = 0.003, ANCOVA

3. Secondary Outcome: Percentage Change in Estimated Glomerular Filtration Rate (eGFR)
Description: eGFR was measured using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation. This value at baseline and 12 months was used to calculate the percentage change by [12 month value-baseline value)/baseline value]*100
Time Frame: Baseline, 12 months
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Pasireotide LAR (SOM230) | Placebo Injection
Number analyzed (Participants) | 29 | 12
percentage of change | -0.3 (14) | -2.2 (17.7)
Statistical Analysis 1: Comparison: Pasireotide LAR (SOM230) vs Placebo Injection; Test type: Superiority; p = 0.79, t-test, 2 sided

4. Secondary Outcome: Percentage Change in Serum Creatinine
Description: Serum creatinine level at baseline and 12 months was used to calculate the percentage change by [12 month value-baseline value)/baseline value]*100
Time Frame: Baseline, 12 months
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Pasireotide LAR (SOM230) | Placebo Injection
Number analyzed (Participants) | 29 | 12
percentage of change | 1.8 (12) | 3.4 (15.6)
Statistical Analysis 1: Comparison: Pasireotide LAR (SOM230) vs Placebo Injection; Test type: Superiority; p = 0.79, t-test, 2 sided

5. Secondary Outcome: Percent Change in Blood Glucose
Description: Blood glucose (mg/dLb) level at baseline and 12 months was used to calculate the percentage change by [12 month value-baseline value)/baseline value]*100
Time Frame: Baseline, 12 months
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Pasireotide LAR (SOM230) | Placebo Injection
Number analyzed (Participants) | 29 | 12
percentage of change | 39 (30) | 2.2 (15.2)
Statistical Analysis 1: Comparison: Pasireotide LAR (SOM230) vs Placebo Injection; Test type: Superiority; p = 0.001, t-test, 2 sided

6. Secondary Outcome: Percentage Change in Hemoglobin A1C
Description: Hemoglobin A1C level at baseline and 12 months was used to calculate the percentage change by [12 month value-baseline value)/baseline value]*100
Time Frame: Baseline, 12 months
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Pasireotide LAR (SOM230) | Placebo Injection
Number analyzed (Participants) | 29 | 12
percentage of change | 18 (11) | 1.6 (3.3)
Statistical Analysis 1: Comparison: Pasireotide LAR (SOM230) vs Placebo Injection; Test type: Superiority; p = 0.001, t-test, 2 sided

7. Secondary Outcome: Percentage Change in Heart Rate
Description: Heart rate, measured in beats per minute (BPM), at baseline and 12 months was used to calculate the percentage change by [12 month value-baseline value)/baseline value]*100
Time Frame: Baseline, 12 months
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Pasireotide LAR (SOM230) | Placebo Injection
Number analyzed (Participants) | 29 | 12
percentage of change | -0.15 (0.2) | -0.1 (0.1)
Statistical Analysis 1: Comparison: Pasireotide LAR (SOM230) vs Placebo Injection; Test type: Superiority; p = 0.73, t-test, 2 sided

8. Secondary Outcome: Change in Quality of Life
Description: Measured using the SF-36 health survey, which consist of eight subscales each scored on a range of 0 to 100 (0=worst imaginable, 100=best imaginable). Change calculated from baseline = 12 month value-baseline value
Time Frame: Baseline, 12 months
Population: Data for 19 participants in the pasireotide LAR (SOM230) group and 9 participants from the placebo injection group was available for analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pasireotide LAR (SOM230) | Placebo Injection
Number analyzed (Participants) | 19 | 9
units on a scale
  Physical functioning | 4.7 (16) | -1 (8)
  Physical role | 7.9 (36) | -3 (38)
  Bodily pain | 5.5 (22) | 7 (12)
  General health | -6.2 (14) | 2 (15)
  Vitality | 4.5 (14) | -2 (17)
  Social functioning | 0.0 (18) | -3 (8)
  Role emotional | 0.0 (22) | 11 (5)
  Mental health | 1.5 (12) | -1.8 (11)
Statistical Analysis 1: Comparison: Pasireotide LAR (SOM230) vs Placebo Injection; Physical functioning; Test type: Superiority; p = 0.31, t-test, 2 sided
Statistical Analysis 2: Comparison: Pasireotide LAR (SOM230) vs Placebo Injection; Physical role; Test type: Superiority; p = 0.48, t-test, 2 sided
Statistical Analysis 3: Comparison: Pasireotide LAR (SOM230) vs Placebo Injection; Bodily pain; Test type: Superiority; p = 0.89, t-test, 2 sided
Statistical Analysis 4: Comparison: Pasireotide LAR (SOM230) vs Placebo Injection; General health; Test type: Superiority; p = 0.18, t-test, 2 sided
Statistical Analysis 5: Comparison: Pasireotide LAR (SOM230) vs Placebo Injection; Vitality; Test type: Superiority; p = 0.28, t-test, 2 sided
Statistical Analysis 6: Comparison: Pasireotide LAR (SOM230) vs Placebo Injection; Social functioning; Test type: Superiority; p = 0.66, t-test, 2 sided
Statistical Analysis 7: Comparison: Pasireotide LAR (SOM230) vs Placebo Injection; Role emotional; Test type: Superiority; p = 0.43, t-test, 2 sided
Statistical Analysis 8: Comparison: Pasireotide LAR (SOM230) vs Placebo Injection; Mental health; Test type: Superiority; p = 0.51, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to 12 months
Arm/Group | Pasireotide LAR (SOM230) | Placebo Injection
All-Cause Mortality (participants affected / at risk) | 0/33 | 1/15
Serious Adverse Events (participants affected / at risk) | 4/33 | 1/15
Other Adverse Events (participants affected / at risk) | 33/33 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pasireotide LAR (SOM230) (N=33) | Placebo Injection (N=15)
Ruptured liver cyst (Hepatobiliary disorders) | 1 (1) | 0 (0)
Elevated alkaline phosphatase (Hepatobiliary disorders) | 1 (1) | 0 (0)
Prolonged QT>480msec (Cardiac disorders) | 1 (1) | 0 (0)
Right upper quadrant pain (General disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (General disorders) | 1 (1) | 0 (0)
Abdominal hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Pasireotide LAR (SOM230) (N=33) | Placebo Injection (N=15)
Hyperglycemia (Metabolism and nutrition disorders) | 26 (26) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 17 (17) | 8 (8)
Dizziness (Nervous system disorders) | 10 (10) | 3 (3)
Pain abdomen (Gastrointestinal disorders) | 11 (11) | 1 (1)
Fatigue (General disorders) | 13 (13) | 3 (3)
Diabetes (Endocrine disorders) | 19/32 (19) | 1 (1)
Nausea (Gastrointestinal disorders) | 9 (9) | 3 (3)
Bradycardia (Cardiac disorders) | 10 (10) | 1 (1)
Alopecia (General disorders) | 9 (9) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-14): https://cdn.clinicaltrials.gov/large-docs/10/NCT01670110/Prot_SAP_000.pdf